CLINICAL TRIAL: NCT05103020
Title: A Randomized, Open-label, Single-center Phase II Study Comparing Conversion Rate to Surgery With Hepatic Arterial Infusion Chemotherapy to Systemic Chemotherapy in Patients With Non Resectable Liver-only Colorectal Metastases
Brief Title: Phase II Study Comparing Conversion Rate to Surgery With Hepatic Arterial Infusion Chemotherapy to Systemic Chemotherapy in Patients With Non Resectable Liver-only Colorectal Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0034
Record Dates: First submitted 2021-10-14; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAI oxaliplatin and systemic FOLFIRI plus targeted therapy (bevacizumab or cetuximab) (Experimental): HAI-oxaliplatin + Systemic FOLFIRI + target agent (bevacizumab or cetuximab)
  Interventions: Drug: intra-arterial oxaliplatin + Systemic FOLFIRI + target agent (bevacizumab or cetuximab) every 2 weeks
- Systemic FOLFIRI plus targeted therapy (bevacizumab or cetuximab) (Active Comparator): IV FOLFIRI+ target agent (bevacizumab or cetuximab)
  Interventions: Drug: IV FOLFIRI+ target agent (bevacizumab or cetuximab) every 2 weeks

INTERVENTIONS:
Drug: intra-arterial oxaliplatin + Systemic FOLFIRI + target agent (bevacizumab or cetuximab) every 2 weeks — Bevacizumab : 5mg/kg IV over 30min, day 1 or Cetuximab : 500 mg/m2 IV over 2-hr, day 1 Oxaliplatin : HAI 100mg/m2 IV over 2-hr, day 1 Leucovorin : 400mg/m2 IV over 2-hr, day 1 5-Fluorouracil : 2400mg/m2 infusion for 46-h Irinotecan : 180mg/m2 IV over 1.5-hr, day 1
  Arms: HAI oxaliplatin and systemic FOLFIRI plus targeted therapy (bevacizumab or cetuximab)
Drug: IV FOLFIRI+ target agent (bevacizumab or cetuximab) every 2 weeks — Bevacizumab : 5mg/kg IV over 30min, day 1 or Cetuximab : 500 mg/m2 IV over 2-hr, day 1 Irinotecan : 180mg/m2 IV over 1.5-hr, day 1 Leucovorin : 400mg/m2, IV over 2-hr, day 1 5-Fluorouracil : 400mg/m2 IV bolus, day 1 5-Fluorouracil : 2400mg/m2, infusion for 46-h
  Arms: Systemic FOLFIRI plus targeted therapy (bevacizumab or cetuximab)

SUMMARY:
Approximately 40% of colorectal cancer patients will develop colorectal liver metastases (CRLM). The most effective approach to increase long-term survival is CRLM complete resection. Unfortunately, only 10 - 15% of CRLM are initially considered resectable. The objective response rates (ORR) after current first-line systemic chemotherapy (sys-CT) regimens range from 40 to 80% and complete resection rates (CRR) range from 25 to 50% in patients with initially unresectable CRLM. When CRLM patients are not amenable to complete resection after induction of sys-CT, ORRs obtained with second-line sys-CT are much lower (between 10 and 30%) and consequently CRRs are also low (< 10%). Hepatic arterial infusion (HAI) oxaliplatin may represent a salvage therapy in patients with CRLM unresectable after one or more sys-CT regimens with ORRs and CRRs up to 60 and 30%, respectively. This study is designed to evaluate the efficacy of an intensification strategy based on HAI oxaliplatin combined with sys-CT as the first-line treatment in patients with unresectable CRLM.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer (CRC), and radiologic or histologic proof of liver metastasis.
2. Unresectability of the CRLM will be confirmed by a centralized multidisciplinary expert panel (composed of surgeons, radiologists, interventional radiologists and medical oncologists). The panel will review the CT scan and MRI of the patients (weekly web conference). Non-resectability criteria (one of the following criteria):

   * Upfront R0/R1 resection of all CRLM (that leaves at least two adequately perfused and drained segments) is not possible
   * Liver metastases in contact with major vessels of the remnant liver which would require resection of the vessel for an R0 resection (i.e., tumor involvement of main portal right and left portal veins, of the three main hepatic veins, or of the retrohepatic vena cava)
3. At least one measurable liver metastasis according to the RECIST v1.1
4. Age ≥18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
6. Life expectancy of at least 3 months
7. Normal liver function International normalized ratio (INR) <1.5 ULN
8. Neutrophils >1500/mm³
9. Platelet >100 x 109/L (transfusion allowed)
10. Hemoglobin >9 g/dL (transfusion allowed)
11. Bilirubin <1.5 times the upper limit of normal values (ULN)
12. Aminotransferases <5 ULN, alkaline phosphatase <5 ULN
13. Calculated creatinine clearance >30 mL/min (Cockcroft and Gault formula)
14. Urine dipstick for proteinuria of less than 1+ is required within 7 days prior to study entry; if urine dipstick is >= 2+ then a 24 hour urine for protein must demonstrate =< 1 gm of protein in 24 hours to allow participation in the study; NOTE: Urinalysis is also acceptable
15. Informed consent signed by the patient or his/her legal representative

Exclusion Criteria:

1. Patient eligible for curative-intent treatment of CRLM (i.e. resection and/or thermoablation), according to the local multidisciplinary team and/or the central review. Definitive anatomical contraindication to complete surgical resection (any of the following criteria):

   * More than two lesions in all liver segments
   * Bilobar liver metastasis and more than three lesions >3 cm in the hepatic lobe the least affected (i.e. the future remnant liver)
   * Bilobar liver metastasis and disease liver extend >50%
2. Extrahepatic tumor disease (except ≤3 lung nodules <10 mm deemed amenable to curative-intent resection/thermoablation and non-resected primary tumor with no or mild symptoms)
3. Major surgical procedure within 28 days prior to study treatment start, or patients who have not fully recovered from major surgery
4. Radiotherapy to target lesion within 4 weeks before the study (A 2-week washout is permitted for palliative radiation.)
5. Has known uncontrolled active CNS metastases and/or carcinomatous meningitis
6. Peripheral neuropathy CTCAE v4.03 ≥ grade 2
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Participants with (A) basal cell carcinoma of skin, (B) squamous cell carcinoma of the skin, (C) low grade thyroid cancer or carcinoma in situ (eg, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy, such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic systemic treatment and is allowed.
9. Uncontrolled hypertension or clinically active cardiovascular disease: for example, cerebrovascular accident or transient ischemic attack, unstable angina, myocardial infarction within 24 weeks prior to randomization. Have symptomatic congestive heart failure (CHF; New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
10. Have significant bleeding disorders, or evidence of bleeding diathesis or coagulopathy
11. Have had a significant bleeding episode from the gastrointestinal (GI) tract or lung
12. Have a history of GI perforation and/or fistula, or intra-abdominal abscess within 24 weeks prior to randomization.
13. Have a history of HNPCC syndrome or polyposis
14. Have experienced any arterial thromboembolic event or ongoing treatment with anticoagulants for therapeutic purpose within 24 weeks prior to randomization.
15. Has a known history of human immunodeficiency virus (HIV) infection
16. Are pregnant or breast feeding. Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to first dose of study treatment. For women of childbearing potential and men, agreement to remain abstinent or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 30 days after the last dose of study drugs. Postmenopausal women is defined that : 1) must have been amenorrheic for at least 12 months, > 50 years old or 2) Age ≤ 50 years old and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range (>40 mIU/mL), 3) prior bilateral oophorectomy
17. Patients who are hypersensitive reaction to experimental drugs
18. Patients who are hypersensitive to CHO cell products or other recombinant or humanized antibodies
19. In case of contraindication of experimental drugs
20. Have any condition (eg, psychological, geographical, or medical) that does not permit compliance with the study and follow-up procedures or suggest that the patient is, in the investigator's opinion, not an appropriate candidate for the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
curative-intent resection rate | Every 4 cycles of chemotherapy (approximately 24 months) (each cycle is 2weeks)
  The primary study objective is to compare the rate of conversion to resectable liver after HAI plus sys-CT and sys-CT alone in colorectal cancer patients with previously untreated and unresectable liver metastases at diagnosis. Randomized patients will receive either chemotherapy combining HAI oxaliplatin plus systemic FOLFIRI and targeted therapy (bevacizumab or cetuximab) or systemic FOLFIRI and targeted therapy (bevacizumab or cetuximab).

SECONDARY OUTCOMES:
Overall survival | Every 8 weeks from date of first treatment until the date of death from any cause, assessed approximately up to 24 months
Progression-free survival | Every 8 weeks from date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed approximately up to 24 months
Toxicity profile | Every 4 weeks from date of first treatment until date of last treatment up to 24 months
  Overall safety profile verified as relevance of adverse events and laboratory abnormality in the study and grades granted based on (USA National Cancer Center) Common Terminology Criteria for Adverse Events such as the type, frequency and severity (CTCAE), v4.0.
Overall response rate (ORR) | Every 8 weeks from date of first treatment until date of last treatment up to 24 months
  Overall objective response rate (ORR) is the best response rate stipulated as complete response (CR) or partial response (PR) (target lesion and tumor response defined according to RECIST guideline version 1.1) and identified as percentage of the confirmed patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dai Hoon Han, M.D, Ph.D, Principal Investigator — Department of Hepatobiliary and Pancreatic Surgery, Yonsei University College of Medicine; Joong Bae Ahn, M.D, Ph.D, Principal Investigator — Division of Medical Oncology, Department of Internal Medicine, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JS, Kim H, Lee SY, Han YD, Han K, Min BS, Kim MD, Won JY, Beom SH, Shin SJ, Kim HS, Han DH, Ahn JB. Hepatic arterial infusion in combination with systemic chemotherapy in patients with hepatic metastasis from colorectal cancer: a randomized phase II study - (NCT05103020) - study protocol. BMC Cancer. 2023 Jul 22;23(1):691. doi: 10.1186/s12885-023-11085-w. PMID 37481515